CLINICAL TRIAL: NCT02133690
Title: Phase III, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Live Attenuated Bovine-Human Rotavirus Reassortant Pentavalent Vaccine (BRV-PV) Against Severe Rotavirus Gastroenteritis in Healthy Indian Infants
Brief Title: A Clinical Trial to Study the Effect and Safety of Rotavirus Vaccine Against Severe Rotavirus Gastroenteritis in Healthy Indian Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Collaborators: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ROTA:03/12
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Rotavirus Gastroenteritis
Keywords: rotavirus; rotavirus vaccine; BRV-PV

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine Arm (Experimental): 3 doses, 4 weeks apart, of Live Attenuated Pentavalent (G1-G2-G3-G4-G9) Human X Bovine Reassortant Rotavirus Vaccine (BRV-PV), at a dosage of ≥ Log10^5.6 fluorescent focus units (FFU)/Serotype/Dose in 2.5 ml of buffered diluent
  Interventions: Biological: Live Attenuated Pentavalent (G1-G2-G3-G4-G9) Human X Bovine Reassortant Rotavirus Vaccine (BRV-PV)
- Placebo group (Placebo Comparator): 3 doses, 4 weeks apart, of Lyophilized minimal essential medium (MEM) + excipients reconstituted in 2.5 ml of buffered diluents
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Live Attenuated Pentavalent (G1-G2-G3-G4-G9) Human X Bovine Reassortant Rotavirus Vaccine (BRV-PV) — Live Attenuated Pentavalent (G1-G2-G3-G4-G9) Human X Bovine Reassortant Rotavirus Vaccine (BRV-PV), at a dosage of ≥ Log10^5.6 fluorescent focus units (FFU)/Serotype/Dose in 2.5 ml of buffered diluent
  Arms: Vaccine Arm
Other: Placebo — Lyophilized minimal essential medium (MEM) + excipients reconstituted in 2.5 ml of buffered diluents
  Arms: Placebo group

SUMMARY:
This is a Phase 3 multicentre, randomized, double blind, placebo-controlled study to determine the effectiveness of the rotavirus vaccine.

DETAILED DESCRIPTION:
The hypothesis is that a three dose series of BRV-PV administered orally to healthy Indian infants, with the initial dose given at 6-8 weeks of age and followed by vaccinations at monthly intervals, will significantly reduce the incidence of severe rotavirus gastroenteritis (SRVGE). Duration of follow-up is until aged 2 years of each enrolled child. The study is powered to detect vaccine efficacy significantly greater than 10% (95% confidence interval lower bound > 10%) if the true vaccine efficacy is 50% or higher.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants as established by medical history and clinical examination before entering the study.
* Age: 6-8 weeks at the time of enrollment.
* Parental ability and willingness to provide informed consent.
* Parent who intends to remain in the area with the child during the study period.

Exclusion Criteria:

* Presence of diarrhea or vomiting in the previous 72 hours or on the day of enrollment (temporary exclusion)
* Presence of fever on the day of enrollment (temporary exclusion).
* Acute disease at the time of enrollment (temporary exclusion)
* Concurrent participation in another clinical trial throughout the entire timeframe for this study.
* Presence of significant malnutrition (weight-for-height z-score <-3SD median) or any systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrine, immunological, dermatological, neurological, cancer or autoimmune disease) as determined by medical history and/or physical examination which would compromise the subject's health or is likely to result in nonconformance to the protocol. History of congenital abdominal disorders, intussusception or abdominal surgery
* Known or suspected impairment of immunological function based on medical history and physical examination.
* Household contact with an immunosuppressed individual or pregnant woman.
* Prior receipt of rotavirus vaccine.
* A known sensitivity or allergy to any components of the study vaccine.
* Major congenital or genetic defect.
* History of persistent diarrhea (defined as diarrhea more than 14 days).
* Participant's parents not able, available or willing to accept active weekly follow-up by the study staff.
* Has received any immunoglobulin therapy and/or blood products since birth or planned administration during the study period.
* History of chronic administration (defined as more than 14 days) of immunosuppressants including corticosteroids. Infants on inhaled or topical steroids may be permitted to participate in the study.
* History of any neurologic disorders or seizures.
* Any medical condition in the parents/infant which, in the judgment of the investigator, would interfere with or serves as a contraindication to protocol adherence or a participant's parents' ability to give informed consent.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7500 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
occurrence of Severe Rotavirus Gastroenteritis | Up to 2 years of age of participants
  Laboratory confirmed cases of severe rotavirus gastroenteritis occurring in infants receiving the complete vaccination regimen occurring from 14 days after the third vaccine dose until 122 cases are accrued, or until all participating infants reach two years of age (per protocol analysis).

SECONDARY OUTCOMES:
Safety | Until completion of 2 years age of participant
  Occurrence of SAE
  * Solicited post-vaccination reactions
  * SAEs
  * Severe AEs
  * Unsolicited AEs
  * Intussusception
  * Death

CONTACTS AND LOCATIONS:
Overall Officials: Prasad Kulkarni, MD, Study Director — Serum Institute of India Pvt. Ltd.
Locations (6):
- India (6):
  - Dr Dinesh Kumar Government Medical College, Jammu Department of Community Medicine, Government Medical College, Jammu, Jammu and Kashmir
  - Kasturba Medical College, Manipal, Manipal, Karnataka
  - KEM Hospital and Research Centre, Pune, Maharashtra
  - Dr. Sushila Nayar School of Public Health ,Mahatma Ghandi School of Medicine, Sewāgrām, Maharashtra
  - Center for Health Research and Development (CHRD) -Society for applied studies (SAS), New Delhi, National Capital Territory of Delhi
  - National Institute of Cholera & Enteric Diseases, Kolkata, West Bengal

REFERENCES:
- [Result] Kulkarni PS, Desai S, Tewari T, Kawade A, Goyal N, Garg BS, Kumar D, Kanungo S, Kamat V, Kang G, Bavdekar A, Babji S, Juvekar S, Manna B, Dutta S, Angurana R, Dewan D, Dharmadhikari A, Zade JK, Dhere RM, Fix A, Power M, Uprety V, Parulekar V, Cho I, Chandola TR, Kedia VK, Raut A, Flores J; SII BRV-PV author group. A randomized Phase III clinical trial to assess the efficacy of a bovine-human reassortant pentavalent rotavirus vaccine in Indian infants. Vaccine. 2017 Oct 27;35(45):6228-6237. doi: 10.1016/j.vaccine.2017.09.014. Epub 2017 Sep 26. PMID 28967523
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5651219/